CLINICAL TRIAL: NCT06525363
Title: Clinical Assessment of Chitosan Nano-particles on Periodontal Problems Post Steroidal Inhalation in Asthmatic Patients: Phase I Trial
Brief Title: Clinical Assessment of Chitosan Nanoparticles on Periodontal Problems Post Steroidal Inhalation in Asthmatic Patients: Phase I Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, associate professor of pharamcy practices, faculaty of pharmacy, Deraya University, Deraya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dental 2024
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Chitosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): chitosan nanoparticles spray 1% w/w twice daily
  Interventions: Drug: Chitosan
- control group (No Intervention): normal healthy hygiene of mouth

INTERVENTIONS:
Drug: Chitosan — chitosan nanoparticles 1%w/w will be formulated in form of spray for oral application twice daily
  Arms: treatment group

SUMMARY:
Periodontal problems management is the most important goals of chronic asthmatic patients that adapted to use steroid inhalation for long time. Gram negative anaerobic bacteria are generally suggested as the primary cause of Periodontal problems and mechanical procedure is the treatment approach, which is performed nonsurgical or surgically. The understanding of the role of bacteria in the initiation and progression of periodontal disease has led to great interest in the use of antibiotics to suppress or eradicate pathogenic macrobiotic. Systemic antibiotics have been used in different forms of periodontal disease treatment. Systemic antibiotics can penetrate soft tissues and may target invasive organisms, can be used to treat multiple sites simultaneously, and may also affect reservoirs of bacterial reinfection such as saliva, the tonsils, and the oral mucosa. However, there may be problems associated with the use of systemic antibiotics such as the development of resistant bacteria, and potential side effects (hypersensitivity reactions, gastrointestinal discomfort, etc.). so in this study we aimed at To evaluate the effect of chitosan nanoparticle spray in management of dental problems in asthmatic patients receiving corticosteroids inhaler that support the growth of bacteria in periodontal area.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-50 years old
* Both sex male and female
* Patients diagnosed as Asthmatic
* Patients treated with corticosteroids inhaler or ( beta2-adrenergic agonist inhaler or nebulizer for their symptoms)

Exclusion Criteria:

* Patients treated with other medication
* Patients not diagnosed as asthmatic
* Comorbidity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Levels of oral Streptococcus mutans | each 3 weeks for 12 weeks
  counting number of of S. mutans will be obtained by culture and be expressed in colony forming units (CFUs)
Plaque Examination | each 3 weeks for 12 weeks
  Plaque is recorded using the plaque index (PI)
The inflammatory status of the gingiva | each 3 weeks for 12 weeks
  recorded using the gingival index (GI)

CONTACTS AND LOCATIONS:
Locations (1):
- Soad A. Mohamad, Minya, Select Region, Egypt

IPD SHARING:
Plan to Share IPD: No